CLINICAL TRIAL: NCT06568718
Title: A Multicenter, Randomized, Parallel, Controlled, Prospective, Open-label Study of the Efficacy and Safety of Longidaze Lyophilisate for Solution for Injections and Rectal Suppositories 3,000 IU in the Combined Treatment of Patients With Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia
Brief Title: Efficacy and Safety of Longidaze in the Treatment of Lower Urinary Tract Symptoms Associated With Benign Prostatic Hyperplasia
Acronym: ADAM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-ADAM-23
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2024-08

CONDITIONS: Lower Urinary Tract Symptoms; Prostatic Hyperplasia
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Longidaze + Tamsulosin (Experimental)
  Interventions: Drug: bovhyaluronidase azoximer; Drug: tamsulosin
- Tamsulosin (Active Comparator)
  Interventions: Drug: tamsulosin

INTERVENTIONS:
Drug: bovhyaluronidase azoximer — Longidaze 3000 IU intramuscularly once every 5 days with a course of 5 injections; Longidaze 3000 IU rectal suppositories once every 3 days with a course of 10 applications; Longidaze 3000 IU rectal suppositories once every 7 days with a course of 10 applications.
  Other Names: Longidaze
  Arms: Longidaze + Tamsulosin
Drug: tamsulosin — Tamsulosin 0.4mg per os every day

SUMMARY:
The goal of this clinical trial is to learn if Longidaze works to treat lower urinary tract symptoms in adult males with benign prostatic hyperplasia. It will also learn about the safety of Longidaze. The main question it aims to answer is:

* Does addition of Longidaze to tamsulosin lower the severity of symptoms assessed by International Prostate Symptom Score?
* What medical problems do participants have under the combined treatment by Longidaze and tamsulosin?

Researchers will compare combined therapy (Longidaze + tamsulosin) with monotherapy (tamsulosin only) to see if the combination works better.

Participants will:

* Take tamsulosin (0.4mg) every day for 130 days
* In combined therapy arm -- make intramuscular injections of Longidaze every 5 days (5 injections); then apply Longidaze rectal suppositories every 3 days (10 applications); then apply Longidaze rectal suppositories every 7 days (10 applications)
* Visit the clinic on day 1, 26±1, 60±1, 130±3 for checkups and tests

ELIGIBILITY:
Inclusion Criteria:

1. Signed Written Informed Consent Form for participation in the study.
2. Male outpatients aged 40 years or older.
3. Presence of lower urinary tract symptoms due to BPH at least 6 months prior to the screening visit.
4. Symptom severity according to the International Prostate Symptom Score (IPSS) ≥ 8 at the screening visit.
5. Negative urethral smear (PCR) test for chlamydia, gonorrhea, trichomoniasis, mycoplasmosis and ureaplasmosis performed no earlier than 1 month prior to study inclusion.
6. Negative blood test (ELISA) for syphilis performed no earlier than 1 month prior to study inclusion.
7. Maximum urine flow rate (Qmax) based on uroflowmetry results during screening is ≥5 ml/sec; residual urine volume during screening is up to 150 ml.
8. Consent to follow the effective methods of contraception specified in the protocol throughout the study.

Exclusion Criteria:

1. History of hypersensitivity to the study drug, background therapy drug or their components or intolerance thereof.
2. Patients who require or do not wish to stop taking drugs prohibited before or during the study.
3. Contraindications to the study therapy at the time of screening: acute infectious diseases; pulmonary hemorrhage and hemoptysis; fresh vitreous hemorrhage.
4. Hematuria, hematological diseases, oncological diseases, chronic heart failure class III-IV according to the New York Heart Association system, diabetes mellitus, chronic renal failure, hypogonadism in the history.
5. Acute prostatitis at the time of screening and/or within 4 weeks before screening.
6. Symptoms of urinary tract infection at the time of screening and/or within 4 weeks before the screening visit.
7. Need for planned surgical treatment of BPH and/or any other concomitant disease within 5 months from the screening visit.
8. History of prostatectomy, transurethral resection and/or other surgical interventions on the prostate gland, bladder or pelvic organs.
9. Neurogenic dysfunction of the bladder, congenital anomalies of the genitourinary system, sclerosis of the bladder neck, bladder diverticula, urolithiasis, bladder cancer or other bladder diseases in the medical history.
10. History of urethral stricture.
11. History of spinal injury.
12. Prostate-specific antigen (PSA) level >4 ng/ml at the screening visit or according to laboratory tests performed no more than 4 weeks before inclusion in the study.
13. History of acute urinary retention.
14. Use of any antibacterial drugs (except topical drugs) within 2 months before the screening visit.
15. Use of any medications for the treatment of LUTS/BPH before the study, including herbal preparations containing extracts of Serenoa repens and Pygeum Africanum.
16. History of orthostatic hypotension.
17. Patients with significant liver dysfunction at the screening visit: total bilirubin >2 ULN, albumin <35 g/L, prothrombin time >3 ULN.
18. Patients with significant renal dysfunction at the screening visit (blood creatinine >2 ULN), and / or patients on dialysis and / or patients with a history of kidney transplant.
19. The patient is scheduled for cataract or glaucoma surgery within 5 months after screening.
20. The presence of sexually transmitted diseases at the time of screening.
21. Patients with positive blood test results for HIV and/or hepatitis B and/or hepatitis C, performed no earlier than 1 month before the screening visit, or at the screening.
22. Decompensated diabetes mellitus (blood glucose and/or HbAc1 grade 3 or higher according to the used CTCAE 4.03 classifier);
23. Severe CNS diseases, including a history of seizures or conditions that may lead to their development; stroke or transient ischemic attack within 12 months before screening; traumatic brain injury or cases of loss of consciousness within 12 months before screening; brain tumor
24. Patients with mental disorders such as psychosis, manic-depressive disorders, chronic depression.
25. Acute or chronic gastric and/or duodenal ulcer at the time of screening.
26. History of alcoholism, drug addiction, drug abuse.
27. Participation in other interventional clinical trials of drugs less than 90 days before the screening visit.
28. Any conditions that, in the opinion of the Investigator, may interfere with the patients participation in the study, compliance with the procedures, or be contrary to his interests, as well as affect the results of the study.
29. Employees of the study center or the Sponsor company, their family members or subjects in dependent relationships.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2024-02-09 (Actual); Study Completion 2024-02-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in IPSS Score on Day 60 and 130 | Day 0, Day 60, Day 130
  Change in symptom severity assessed by the patient using the International Prostate Symptom Score (IPSS) relative to baseline on days 60 and 130 of therapy. IPSS score ranges from 0 to 35 with higher score representing more severe symptoms.

SECONDARY OUTCOMES:
Change from Baseline in IPSS Score on Day 26 | Day 0, Day 26
  Change in symptom severity assessed by the patient using the International Prostate Symptom Score (IPSS) relative to baseline on day 26 of therapy. IPSS score ranges from 0 to 35 with higher score representing more severe symptoms.
Change from Baseline in Qmax | Day 0, Day 26, Day 60, Day 130
  Change in maximum urine flow rate (Qmax) according to uroflowmetry relative to baseline
Change from Baseline in Prostate Volume | Day 0, Day 26, Day 60, Day 130
  Change in prostate volume relative to baseline
Number of Participants with 4 Points and/or 25% Decrease in IPSS Score | Day 0, Day 26, Day 60, Day 130
  Proportion of patients showing a decrease in symptom severity as assessed by the IPSS questionnaire by 4 or more points and/or by 25% from the baseline.
Change from Baseline in IPSS QoL Score | Day 0, Day 26, Day 60, Day 130
  Change in quality of life (QoL) assessed by the patient using the International Prostate Symptom Score (IPSS, QoL domain) relative to baseline. IPSS QoL score ranges from 0 ("delighted") to 6 ("terrible").
Change from Baseline in IPSS-V Score | Day 0, Day 26, Day 60, Day 130
  Change in voiding symptom severity assessed by the patient using the IPSS questionnaire (IPSS-V subscore) relative to baseline. IPSS-V score ranges from 0 to 20 with higher score representing more severe symptoms.
Change from Baseline in IPSS-S Score | Day 0, Day 26, Day 60, Day 130
  Change in storage symptom severity assessed by the patient using the IPSS questionnaire (IPSS-S subscore) relative to baseline. IPSS-S score ranges from 0 to 15 with higher score representing more severe symptoms.
Change from Baseline in Residual Urine Volume | Day 0, Day 26, Day 60, Day 130
  Change in residual urine volume based on ultrasound data relative to baseline
Change from Baseline in NIH-CPSI Score | Day 0, Day 26, Day 60, Day 130
  Change in symptom severity according to the NIH Chronic Prostatitis Symptom index (NIH-CPSI) questionnaire relative to the baseline

OTHER OUTCOMES:
Number of Participants with Treatment-Related Adverse Events | From enrollment to the end of treatment on Day 130
  Safety assessment based on laboratory test data, evaluation of the vital signs, physical examination, and registration of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel I. Rasner, Principal Investigator — University Clinic of the Scientific and Educational Institute of Clinical Medicine named after N.A. Semashko
Locations (3):
- Russia (3):
  - LLC "Krasnodar Medical and Biological Center", Krasnodar
  - First Saint Petersburg State Medical University named after academician I.P. Pavlov, Saint Petersburg
  - LLC "Clinic of Modern Medicine of Dr. Bogorodskaya", Yaroslavl

IPD SHARING:
Plan to Share IPD: No